CLINICAL TRIAL: NCT01801085
Title: The Impact of Nursing and Pharmacy Care Between Xeloda® and 5-Fluoruracil Regimens in the Management of Colorectal Cancer (CRC) in Hong Kong
Brief Title: Nursing and Pharmacy Time for Delivering Xeloda® Versus 5-Fluoruracil Regimens
Status: Terminated | Type: Observational
Why Stopped: Slow recruitment pace
Sponsor: Vivian Wing Yan Lee (Other)
Collaborators: Hoffmann-La Roche (Industry); Queen Elizabeth Hospital, Hong Kong (Other); Princess Margaret Hospital, Hong Kong (Other Government)
Responsible Party: Sponsor-Investigator, Vivian Wing Yan Lee, Associate Professor, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Other Study IDs: Roche-TR116581; TR116581VLKZ002 (Other: CUHK)
Record Dates: First submitted 2012-09-05; First posted 2013-02-28 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-02

CONDITIONS: Colorectal Cancer
Keywords: Time-and-Motion; Neoplasm; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FOLFOX4: Leucovorin 200 mg/m2 iv over 2 hrs before 5-FU, d1 and 2 5-FU 400 mg/m2 iv bolus and then 600 mg/m2 iv over 22 hrs, d 1 and d2 Oxaliplatin (Eloxatin) 85 mg/m2 iv d1 Q2w x 12 cycles
- XELOX: Capecitabine (Xeloda) 1000 mg/m2 po bid x 14 days Oxaliplatin (Eloxatin) 130 mg/m2 iv over 2 hrs d1 Q3w x 8 cycles

SUMMARY:
This is a prospective time-and-motion study to document and compare the time used in preparation, dispensing and administration for capecitabine/oxaliplatin (XELOX) versus IV 5-FU/leucovorin/oxaliplatin (FOLFOX4) regimens in colorectal cancer (CRC) patients.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second most common cause of cancer-related death in Hong Kong. The traditional chemotherapy for CRC remains on intravenous (IV) fluorouracil (5-FU) based regimens with the response rates of 10-20% and a median survival of approximately one year. Recent years, oral chemotherapy has a more practical and economic advantages over IV regimen. It is understandable that patients prefer oral regimens as long as the clinical efficacy is maintained. Oral treatment strategy preserves quality of life for CRC patients. In a previous cost-minimization study conducted in Hong Kong, it was demonstrated that capecitabine was more cost-effective than 5-FU plus oxaliplatin assuming they had equal clinical efficacy. Not only is capecitabine more cost-effective, it may also have additional cost saving in the nursing and pharmacy time . It is because a significant amount of time can be saved in both nursing and pharmacy for the preparation and administration of IV chemotherapy. In the UK, it was demonstrated that capecitabine required less pharmacy and administration time per cycle than 5-FU based IV chemotherapy. However, there is a lack of local data to demonstrate the impact of pharmacy and nursing care utilizing capecitabine comparing to traditional IV chemotherapy in CRC patients of Hong Kong.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* Diagnosed with CRC and prescribed with either XELOX for FOLFOX4 chemotherapy treatment

Exclusion Criteria:

* Patients less than 18 years of age
* Persons related unequally to investigators
* Patients who are mentally/cognitively disabled
* Patients who refuse to give consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Colorectal patients who were newly prescribed to receive either the XELOX or the FOLOFX4 chemotherapy regimen will be identified from the colorectal clinic.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2011-10; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Composite preparation, dispensing and administration time | Up to 6 months after the initiation of chemotherapy
  Composite time is measured via real-time recording. Total length of the said time points are to be recorded using a stop-watch and the sum is tabulated in the end.

SECONDARY OUTCOMES:
Capital item utilization (hospital bed and infusion pump) | Up to 6 months after the initiation of chemotherapy
  Capital item utilization is measured as the amount of time each healthcare resource is used and the associated cost for usage.

CONTACTS AND LOCATIONS:
Overall Officials: Vivian WY Lee, PharmD, Principal Investigator — CUHK
Locations (2):
- Hong Kong (2):
  - Princess Margaret Hospital, Kowloon
  - Queen Elizabeth Hospital, Kowloon